CLINICAL TRIAL: NCT04304963
Title: Hypo-METRICS: Hypoglycaemia - Measurement, ThResholds and ImpaCtS A Clinical Study to Determine the Optimal Threshold and Duration of Low Interstitial Glucose Events That Have an Impact on Patient Experienced Hypoglycaemia, Quality of Life and Health Economic Outcomes.
Brief Title: Hypo-METRICS: Hypoglycaemia - Measurement, ThResholds and ImpaCtS
Acronym: Hypo-METRICS
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: University of Southern Denmark (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Ninewells Hospital (Other); Radboud University Medical Center (Other); Nordsjaellands Hospital (Other); Medical University of Graz (Other); University Hospital, Montpellier (Other); Innovative Medicines Initiative (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); Juvenile Diabetes Research Foundation (Other); International Diabetes Federation (Other); Novo Nordisk A/S (Industry); Abbott Diabetes Care (Industry); Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: 259415
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hypoglycemia; Hypoglycemia Unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T1DM and intact awareness of hypoglycaemia: 200 participants with T1DM and intact awareness of hypoglycaemia
  Interventions: Other: NO intervention - observational study
- T1Dm and impaired awareness of hypoglycaemia: 50 participants with T1Dm and impaired awareness of hypoglycaemia
  Interventions: Other: NO intervention - observational study
- insulin treated T2DM: 350 participants with insulin treated T2DM ( > 1 injections / day)
  Interventions: Other: NO intervention - observational study

INTERVENTIONS:
Other: NO intervention - observational study — NO intervention - observational study

SUMMARY:
Hypoglycaemia or low blood glucose, and its fear are major barriers to achieving optimal glucose control. New technology, such as continuous glucose monitors (CGM), help to better identify hypoglycaemia and develop strategies to avoid it. These devices measure glucose in the skin, rather than in the blood, and provide information not only on how low glucose is, but also for how long. Recent studies showed that over half of episodes of low glucose with these systems are not recognised by people with diabetes, and even people without diabetes have sensor values that are below the current thresholds for hypoglycaemia [ low blood glucose] that we measure with traditional monitors.

In this study, the investigators will evaluate the impact of symptomatic as well as asymptomatic episodes of low sensor glucose on a variety of clinical, patient-related and health economic outcomes such as mood, quality of sleep and productivity. The investigators will test different levels and durations of low sensor glucose to identify the one that best matches episodes that are symptomatic to best define hypoglycaemia using these systems.

The investigators will also look at factors that influence this such as sleep or activity as well as diabetes management behaviours (such as insulin dosing, carb counting, etc). At the end of this study, the investigators will be able to provide a better definition of clinically relevant low sensor glucose readings that will help inform clinical as well as academic interpretation of CGM data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 85 years
2. HbA1c 5 - 10% [31 - 86 mmol/mol]
3. Confirmed diagnosis of type 1 or type 2 diabetes
4. Using > 1 injection of insulin / day or insulin pump.
5. Ability to provide written informed consent
6. Performing regular SMBG [ > 1 / day on a 4-week download] . For those using flash or continuous glucose monitoring, this should be used at least 70% of the time.
7. At least 1 episode of hypoglycaemia [ either biochemical or symptomatic] in the last month
8. On stable therapy for at least 3 months.
9. Willing to complete study procedures including wearing the Fitbit and CGM devices and completing the EMA questionnaires on the uMotif app three times a day for 10 weeks ( we expect minimum 80% data completeness)

Exclusion Criteria:

1. Concurrent conditions that can affect glucose readings [renal impairment GFR < 30 ml/min, hepatic impairment, untreated adrenal or thyroid insufficiency, as judged by the investigator.
2. Severe cognitive impairment or psychological illness that can impair performance of EMA tasks, visual impairment that will preclude use of the EMA or sensors.
3. Severe psychiatric / psychological illness including extreme fear of hypo- or hyper- glycaemia ( in the opinion of the investigator)
4. Pregnant or plans for pregnancy in the next 6 months
5. Use of automated insulin delivery systems such as closed loop or automated threshold suspend or predictive low glucose suspend insulin pumps.
6. Known allergies to adhesives required for the CGM systems
7. People who work regular night shifts
8. Any other condition which in the opinion of the study team would impair their ability to complete the study

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 600 participants will be recruited in the following categories.
  * Type 1 diabetes with intact awareness of hypoglycaemia [ Gold score < 3]; a maximum of 50% will be using flash or continuous glucose monitoring [ n = 200 ]
  * Type 1 diabetes with impaired awareness of hypoglycaemia [ gold score > 4 ];[n=50] a maximum of 50% will be using flash or continuous glucose monitoring
  * Type 2 diabetes on > 1 injections; a minimum of 25% of these participants will be over 60 years of age; a maximum of 50% will be using flash or continuous glucose monitoring. [n=350]
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
LIG optimum detection of hypoglycemia | week 10
  To determine the Low Interstitial Glucose (LIG) parameters that have the optimum performance for detection and identification of patient-reported-hypoglycemia (PRH); 〖LIG〗_PRH (h_opt,t_opt).

SECONDARY OUTCOMES:
Secondary outcome 1 | week 10
  To evaluate the impact of symptomatic and asymptomatic hypoglycaemia on different domains of Quality of Life (QoL) and health economic variables measured by a bespoke mobile phone application.
  We will use the definition of LIG identified in the primary objective, 〖LIG〗_PRH (h_opt,t_opt), to evaluate the impact of symptomatic and asymptomatic hypoglycaemia on various outcome variables. To do this, we will divide the days into one of 4 categories LIG-PRH- :no hypoglycaemia LIG+PRH- :asymptomatic biochemical hypoglycaemia ( CGM false positive) LIG+PRH+ :symptomatic biochemical hypoglycaemia LIG-PRH+ :symptomatic without biochemical hypoglycaemia (CGM false negative) We will then compare the scores in different domains collected on the app ( eg reported mood, quality of sleep, alertness, productivity, time off work) between the 4 categories.
Secondary outcome 2 | week 10
  To evaluate the impact of adding co-variates such as change of glucose for 30 minutes prior to the event and area under the curve to the threshold and duration parameters to see if this can improve the sensitivity and specificity of 〖LIG〗_PRH (h_opt,t_opt),
Secondary outcome 3 | week 10
  To evaluate the impact on these optimal parameters [〖LIG〗_PRH (h_opt,t_opt ] on Type of diabetes ( Type 1 with normal awareness, Type 2, Type 1 with impaired awareness) Awake vs sleeping ( as determined by Fitbit) Usual Mode of glucose monitoring (SMBG vs Flash vs CGM) Rate of 〖LIG〗_PRH during the study
Secondary outcome 4 | week 10
  To evaluate the impact of the rate of 〖LIG〗_PRH over the whole study duration on Rate of Patient reported hypoglycaemia ( non-severe) Rate of severe hypoglycaemia Overall EQ-5D-5L scores WPAI ( productivity) PROMIS - (sleep quality) Hypo fear scores Baseline C-peptide levels
Secondary outcome 5 | week 10
  To determine the parameters (threshold and duration) of low interstitial glucose (LIG) that best identify a pre-specified reduction/ change in QoL. [ 0.07 reduction in EQ-5D-5L] 〖LIG〗_(EQ-5D) (h_opt,t_opt).
Secondary outcome 6 | week 10
  To determine the parameters ( threshold and duration) of low interstitial glucose (LIG) that best identify a pre-specified health economic outcome. [1.5 hour loss of effective work/ activity] 〖LIG〗_productivity (h_opt,t_opt).
Secondary outcome 7 | week 10
  Determining the predictors of 〖LIG〗_PRH by looking at variables such as mean glucose, variability, activity (step count and intensity).
Secondary outcome 8 | week 10
  We will evaluate the impact of activity ( step count) on the risk of 〖LIG〗_PRH the following night. A generalized linear mixed models (GLMM) with step count as the independent variable and the rate of LIG_PRH as the response variable will address this research question
Secondary outcome 9 | week 10
  We will try to understand some of the causes of hypoglycaemia. To do this we will look at the 4 hours prior to every available 〖LIG〗_PRH (h_opt,t_opt) and PRH and describe the category of events (if also insulin data is available) by classifying them into those with Bolus within range [ < 10 mmol/l] within 4 hours Bolus and correction [ > 10 mmol/l ] within 4 hours No bolus within 4 hours Activity [ as identified by the Fitbit charge 3] within 2 hours.
Secondary outcome 10 | week 10
  Evaluating the effect of personality (assessed by DS-14) on number and severity of hypoglycaemia and the effect of hypoglycaemia on quality of life measures

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martine-Edith G, Zaremba N, Divilly P, Soholm U, Broadley M, Baumann PM, Mahmoudi Z, Gomes M, Ali N, Abbink EJ, de Galan B, Brosen J, Pedersen-Bjergaard U, Vaag AA, McCrimmon RJ, Renard E, Heller S, Evans M, Cigler M, Mader JK, Amiel SA, Speight J, Pouwer F, Choudhary P. Associations Between Hypoglycemia Awareness Status and Symptoms of Hypoglycemia Among Adults with Type 1 or Insulin-Treated Type 2 Diabetes Using the Hypo-METRICS Smartphone Application. Diabetes Technol Ther. 2024 Aug;26(8):566-574. doi: 10.1089/dia.2023.0596. Epub 2024 Apr 12. PMID 38512385
- [Derived] Martine-Edith G, Divilly P, Zaremba N, Soholm U, Broadley M, Baumann PM, Mahmoudi Z, Gomes M, Ali N, Abbink EJ, de Galan B, Brosen J, Pedersen-Bjergaard U, Vaag AA, McCrimmon RJ, Renard E, Heller S, Evans M, Cigler M, Mader JK, Speight J, Pouwer F, Amiel SA, Choudhary P, Hypo-Resolve FT. A Comparison of the Rates of Clock-Based Nocturnal Hypoglycemia and Hypoglycemia While Asleep Among People Living with Diabetes: Findings from the Hypo-METRICS Study. Diabetes Technol Ther. 2024 Jul;26(7):433-441. doi: 10.1089/dia.2023.0522. Epub 2024 Apr 17. PMID 38386436
- [Derived] Divilly P, Zaremba N, Mahmoudi Z, Soholm U, Pollard DJ, Broadley M, Abbink EJ, de Galan B, Pedersen-Bjergaard U, Renard E, Evans M, Speight J, Brennan A, McCrimmon RJ, Mullenborn M, Heller S, Seibold A, Mader JK, Amiel SA, Pouwer F, Choudhary P; Hypo-RESOLVE Consortium. Hypo-METRICS: Hypoglycaemia-MEasurement, ThResholds and ImpaCtS-A multi-country clinical study to define the optimal threshold and duration of sensor-detected hypoglycaemia that impact the experience of hypoglycaemia, quality of life and health economic outcomes: The study protocol. Diabet Med. 2022 Sep;39(9):e14892. doi: 10.1111/dme.14892. Epub 2022 Jun 22. PMID 35633291
- [Derived] Soholm U, Broadley M, Zaremba N, Divilly P, Nefs G, Mahmoudi Z, de Galan B, Pedersen-Bjergaard U, Brennan A, Pollard DJ, McCrimmon RJ, A Amiel S, Hendrieckx C, Speight J, Choudhary P, Pouwer F; Hypo-RESOLVE Consortium. Investigating the day-to-day impact of hypoglycaemia in adults with type 1 or type 2 diabetes: design and validation protocol of the Hypo-METRICS application. BMJ Open. 2022 Feb 1;12(2):e051651. doi: 10.1136/bmjopen-2021-051651. PMID 35105572